CLINICAL TRIAL: NCT05297578
Title: A Phase 2, Randomized, Observer-Blind, Dose-Finding, Controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 24-Valent Pneumococcal Conjugate Vaccine (VAX-24) in Healthy Adults 65 Years and Older
Brief Title: Safety, Tolerability, and Immunogenicity Study of a 24-Valent Pneumococcal Conjugate Vaccine (VAX-24) in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX24-102
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VAX-24 Low Dose (Experimental): Participants will receive a single dose of VAX-24 1.1 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24-Valent Pneumococcal Conjugate Vaccine
- VAX-24 Mid Dose (Experimental): Participants will receive a single dose of VAX-24 2.2 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24-Valent Pneumococcal Conjugate Vaccine
- VAX-24 Mixed Dose (Experimental): Participants will receive a single dose of VAX-24 2.2 mcg/4.4 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24-Valent Pneumococcal Conjugate Vaccine
- PCV20 (Active Comparator): Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  Interventions: Biological: Pneumococcal 20-valent Conjugate Vaccine

INTERVENTIONS:
Biological: 24-Valent Pneumococcal Conjugate Vaccine — 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
  Arms: VAX-24 Low Dose; VAX-24 Mid Dose; VAX-24 Mixed Dose
Biological: Pneumococcal 20-valent Conjugate Vaccine — 0.5 ml dose of Prevnar 20 will be administered into the deltoid muscle at Day 1
  Other Names: Prevnar 20, PCV20
  Arms: PCV20

SUMMARY:
The objective of the study is to evaluate the safety and tolerability of a single injection of VAX-24 at 3 dose levels compared to Prevnar 20™ (PCV20) in adults 65 years of age and older.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and tolerability of a single injection of VAX-24 at 3 dose levels (Low: 1.1 mcg; Mid: 2.2 mcg; or Mixed: 2.2/4.4 mcg) compared to Prevnar 20™ (PCV20) in adults 65 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 65 or older.
* Able and willing to complete the informed consent process.
* Available for clinical follow-up through the last study visit at 6 months after the study vaccination.
* In good general health as determined by medical history, vital signs, physical examination, and clinical judgment of the investigator. Preexisting medical conditions must be stable as defined by no change in treatment at least 6 weeks prior to study participation.
* Willing to have blood samples collected, stored indefinitely, and used for research purposes.
* Able to provide proof of identity to the satisfaction of the study staff completing the enrollment process.

Exclusion Criteria:

* Previous pneumococcal disease (either confirmed or by self-reporting).
* Previous receipt of a licensed or investigational pneumococcal vaccine.
* Receipt of any investigational study product within 30 days prior to enrollment into the study, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
* Planned or actual administration of any licensed vaccine during the period starting 30 days before enrollment into the study through Day 29.
* Physical examination indicating any clinically significant medical condition.
* Body Temperature > 38.0°C (> 100.4°F) or acute illness within 3 days prior to study vaccination (subject may be rescheduled).
* Previous or existing diagnosis of HIV, Hepatitis B or Hepatitis C.
* History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular injections or blood draws.
* Any other chronic or clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety or rights of the subject or confound evaluation of the study vaccine.
* Any medical, psychiatric, or social condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
* Received blood or blood product (including Immune Globulin IV) within 90 days prior to enrollment into the study.
* Received systemic corticosteroids for ≥ 14 consecutive days and has not completed treatment ≤30 days prior to enrollment into the study.
* Receiving immunosuppressive therapy.
* History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 207 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Vaxcyte, Inc.
Locations (20):
- United States (20):
  - Accel Research Sites-Birmingham Clinical Research Unit, Birmingham, Alabama
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - CenExel RCA, Hollywood, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - AMR Newton, formerly Heartland Research Associates, Newton, Kansas
  - AMR Wichita West, Wichita, Kansas
  - AMR New Orleans, New Orleans, Louisiana
  - Healthcare Research Network, Hazelwood, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Accellacare of Rocky Mount, Rocky Mount, North Carolina
  - Meridian Clinical Research, Cincinnati, Ohio
  - Accellacare of Charleston, Mt. Pleasant, South Carolina
  - Coastal Carolina Research, North Charleston, South Carolina
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - CenExel JBR Clinical Research, Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.

REFERENCES:
- [Result] Wassil J, Sisti M, Fairman J, Rankin B, Clark J, Bennett S, Johnson D, Migone TS, Nguyen K, Paschenko A, Sauer P, Iki S, Hanson ME, Simon JK. A phase 2, randomized, blinded, dose-finding, controlled clinical trial to evaluate the safety, tolerability, and immunogenicity of a 24-valent pneumococcal conjugate vaccine (VAX-24) in healthy adults 65 years and older. Vaccine. 2024 Nov 14;42(25):126124. doi: 10.1016/j.vaccine.2024.07.025. Epub 2024 Jul 17. PMID 39025698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 230 participants were screened; 21 did not meet eligibility criteria and 2 were excluded for other reasons. 1 participant was randomized to VAX-24 2.2 mcg but was administered and included in the analysis for VAX-24 2.2/4.4 mcg dose. 1 participant in the PCV20 group was lost to follow up at day 1 without any solicited or unsolicited AEs collected. A 66-year-old male did not finish due to sudden cardiac death not considered related to vaccine due to risk factors of hypertension and BMI=47.4
Period: Overall Study
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Started | 52 | 52 | 52 | 51
Safety Population (The Safety Population is defined as all subjects in the Exposed Population who provided safety assessment data. One subject was excluded from the safety population because they were lost to follow up on Day 1 without any solicited or unsolicited AEs collected.) | 52 | 52 | 52 | 50
Immunogenicity Evaluable Population (The Immunogenicity Evaluable Population includes all subjects in the Exposed Population who had no major protocol deviation that would impact immunogenicity assessment or other reason to be excluded as defined prior to unblinding or analysis, who had not received a prohibited medication or vaccine, and who provided evaluable serum sample results for baseline and Day 29 within the required protocol time frames.) | 48 | 48 | 47 | 45
Completed | 51 | 50 | 49 | 50
Not Completed | 1 | 2 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- PCV20Group 4: Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  Pneumococcal 20-valent Conjugate Vaccine: 0.5 ml dose of Prevnar 20 will be administered into the deltoid muscle at Day 1
- Total: Total of all reporting groups
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4 | Total
Number analyzed (Participants) | 52 | 52 | 52 | 51 | 207
Age, Continuous [Median (Full Range); unit: Years] | 67.5 [65 to 80] | 66.5 [65 to 79] | 67.0 [65 to 88] | 67.0 [65 to 80] | 67.0 [65 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 37 | 31 | 140
  Male | 14 | 18 | 15 | 20 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 5 | 8 | 25
  Not Hispanic or Latino | 44 | 43 | 46 | 41 | 174
  Unknown or Not Reported | 3 | 2 | 1 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 10 | 14 | 14 | 45
  White | 44 | 41 | 37 | 36 | 158
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 165.5 [157.5 to 171.8] | 166.6 [160.5 to 172.7] | 167.6 [162.6 to 172.7] | 166.4 [162.5 to 175.0] | 166.6 [161.3 to 172.7]
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 75.05 [68.04 to 88.68] | 80.36 [70.09 to 98.80] | 86.11 [69.04 to 95.73] | 81.00 [68.49 to 98.60] | 80.30 [68.95 to 95.30]
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 27.42 [25.08 to 31.47] | 28.98 [25.97 to 35.23] | 29.48 [25.65 to 34.37] | 28.99 [24.68 to 33.97] | 28.82 [25.28 to 33.97]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Local Reactions Within 7 Days After Vaccination
Description: Solicited local reactions included redness/erythema, swelling/induration, and pain at injection site
Time Frame: 7 days after vaccination
Population: Safety population, defined as all participants exposed to study vaccine
Measure: Number; unit: percentage of participants
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 52 | 51 | 53 | 50
percentage of participants
  Any solicited local AE (any grade) | 42.3 | 62.7 | 37.7 | 48.0
  Pain (Local-any grade) | 38.5 | 62.7 | 37.7 | 48.0
  Erythema (redness) at the injection site (any grade) | 3.8 | 3.9 | 3.8 | 10.0
  Edema (swelling) at the injection site (any grade) | 5.8 | 2.0 | 3.8 | 6.0

2. Primary Outcome: Percentage of Participants Reporting Solicited Systemic Events Within 7 Days After Vaccination
Description: Solicited systemic reactions include fever, headache, fatigue, muscle pain, and joint pain within 7 days of vaccination
Time Frame: 7 days after vaccination
Population: Safety population, defined as all participants exposed to study vaccine
Measure: Number; unit: Percentage of participants
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 52 | 51 | 53 | 50
Percentage of participants
  Any solicited systemic AE (any grade) | 34.6 | 41.2 | 28.3 | 44.0
  Fever (any grade) | 0 | 0 | 0 | 0
  Fatigue (any grade) | 26.9 | 31.4 | 15.1 | 14.0
  Headache (any grade) | 17.3 | 11.8 | 11.3 | 16.0
  Muscle Pain (any grade) | 19.2 | 27.5 | 17.0 | 32.0
  Joint pain (any grade) | 9.6 | 11.8 | 5.7 | 4.0

3. Primary Outcome: Percentage of Subjects Reporting Unsolicited Adverse Events Within 1 Month After Vaccination
Description: Percentage of participants with at least one Treatment Emergent Adverse Event (unsolicited AEs and SAEs)
Time Frame: 1 month after vaccination
Population: Safety population. defined as all participants exposed to study vaccine
Measure: Number; unit: Percentage of participants
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 52 | 51 | 53 | 50
Percentage of participants | 11.5 | 7.8 | 5.7 | 16.0

4. Primary Outcome: Percentage of Participants Reporting SAEs and New Onset of Chronic Illnesses (NOCIs)
Description: Percentage of participants with serious adverse events (SAEs) and new onset of chronic illness (NOCIs)
Time Frame: 6 months after vaccination
Population: Safety population, defined as all participants exposed to study vaccine
Measure: Number; unit: Percentage of participants
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 52 | 51 | 53 | 50
Percentage of participants
  Participants with at least 1 SAE | 1.9 | 2.0 | 1.9 | 0.0
  Participants with at least 1 NOCI | 1.9 | 2.0 | 1.9 | 0.0

5. Secondary Outcome: VAX-24 Pneumococcal Serotype-specific Opsonophagocytic Assay (OPA) Geometric Mean Titer (GMTs)
Description: The change from baseline to 1 month post-vaccination in the immune response directed against each of the 24 serotypes was evaluated by measuring serotype-specific functional antibody responses with an opsonophagocytic (OPA) assay that assesses the functional capacity of pneumococcal antibodies.
Time Frame: 1 month after vaccination
Population: Immunogenicity Evaluable Populations, defined as participants in the exposed population with no major protocol deviation that impacted immunogenicity assessment and provided evaluable serum sample results for baseline, the relevant post-vaccination time points, and within the required time frames.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 48 | 47 | 48 | 45
Titer
  1: number analyzed (Participants) | 47 | 47 | 48 | 45
  1 | 288.67 [162.84 to 511.76] | 284.55 [160.15 to 505.57] | 135.10 [75.44 to 241.92] | 182.60 [100.41 to 332.05]
  2 | 1224.83 [824.49 to 1819.55] | 1865.97 [1248.74 to 2788.31] | 1060.68 [703.20 to 1599.89] | 81.26 [53.50 to 123.41]
  3 | 252.56 [176.21 to 361.98] | 311.14 [215.93 to 448.34] | 350.55 [242.06 to 507.66] | 342.86 [234.51 to 501.29]
  4 | 1386.27 [854.33 to 2249.42] | 1375.38 [841.57 to 2247.81] | 1472.75 [895.08 to 2423.25] | 1031.62 [618.98 to 1719.34]
  5 | 340.10 [194.28 to 595.39] | 459.02 [260.04 to 810.25] | 240.64 [135.27 to 428.12] | 390.30 [216.16 to 704.75]
  6A | 1672.35 [841.11 to 3325.09] | 3678.45 [1831.34 to 7388.59] | 2492.54 [1229.08 to 5054.79] | 1877.87 [909.27 to 3878.26]
  6B | 1889.61 [1008.38 to 3540.94] | 2736.64 [1446.86 to 5176.17] | 2827.09 [1481.63 to 5394.35] | 2132.92 [1094.3 to 4157.19]
  7F | 2738.72 [1786.47 to 4198.55] | 2884.67 [1869.80 to 4450.37] | 3725.68 [2400.58 to 5782.22] | 3189.78 [2032.14 to 5006.89]
  8: number analyzed (Participants) | 47 | 47 | 48 | 45
  8 | 1789.95 [1161.06 to 2759.48] | 1970.88 [1273.06 to 3051.21] | 1450.17 [925.72 to 2271.74] | 1498.73 [951.60 to 2360.43]
  9N | 7559.19 [5373.89 to 10633.16] | 7451.59 [5281.82 to 10512.70] | 7295.23 [5120.33 to 10393.93] | 1673.49 [1159.81 to 2414.69]
  9V: number analyzed (Participants) | 48 | 46 | 48 | 45
  9V | 927.63 [519.95 to 1654.98] | 1601.84 [882.94 to 2906.09] | 1858.57 [1024.51 to 3371.61] | 972.10 [526.85 to 1793.63]
  10A | 2544.55 [1497.94 to 4322.45] | 2921.81 [1707.58 to 4999.43] | 2484.44 [1422.17 to 4340.17] | 2490.76 [1425.51 to 4352.07]
  11A: number analyzed (Participants) | 48 | 46 | 48 | 45
  11A | 879.43 [670.80 to 1152.96] | 1068.11 [811.06 to 1406.63] | 1072.92 [811.97 to 1417.72] | 814.61 [610.77 to 1086.49]
  12F | 1060.55 [561.14 to 2004.41] | 1153.52 [604.61 to 2200.78] | 1233.96 [641.05 to 2375.26] | 718.93 [367.24 to 1407.42]
  14: number analyzed (Participants) | 48 | 46 | 48 | 45
  14 | 1972.20 [1252.37 to 3105.78] | 3253.68 [2046.65 to 5172.55] | 1607.64 [1004.25 to 2573.57] | 2491.35 [1530.09 to 4056.51]
  15B: number analyzed (Participants) | 48 | 46 | 48 | 45
  15B | 1964.60 [1099.88 to 3509.16] | 1504.58 [828.17 to 2733.45] | 1489.75 [815.60 to 2721.12] | 1759.25 [946.23 to 3270.81]
  17F | 2010.33 [1448.91 to 2789.27] | 2035.09 [1462.74 to 2831.38] | 1979.30 [1413.38 to 2771.81] | 267.63 [187.62 to 381.76]
  18C | 1553.59 [963.38 to 2505.39] | 2237.89 [1377.93 to 3634.56] | 2894.88 [1770.60 to 4733.03] | 1327.56 [801.76 to 2198.19]
  19A | 3608.79 [2475.63 to 5260.62] | 5805.66 [3960.51 to 8510.44] | 5124.99 [3477.83 to 7552.27] | 3808.09 [2558.49 to 5667.99]
  19F | 1211.40 [795.46 to 1844.84] | 1305.32 [851.81 to 2000.29] | 1723.29 [1117.99 to 2656.34] | 854.85 [548.44 to 1332.47]
  20B | 6871.60 [4184.11 to 11285.29] | 7368.09 [4455.60 to 12184.42] | 6621.65 [3975.31 to 11029.64] | 75.74 [44.06 to 130.19]
  22F | 3326.80 [2010.16 to 5505.82] | 6107.92 [3663.16 to 10184.29] | 4248.38 [2530.07 to 7133.68] | 8596.62 [5051.71 to 14629.07]
  23F | 808.78 [410.58 to 1593.16] | 823.11 [413.68 to 1637.74] | 1182.95 [588.94 to 2376.10] | 630.71 [308.41 to 1289.83]
  33F: number analyzed (Participants) | 48 | 46 | 48 | 45
  33F | 8681.95 [5543.21 to 13597.95] | 11868.64 [7495.14 to 18794.13] | 10621.27 [6694.23 to 16852.03] | 9994.41 [6225.25 to 16045.67]

6. Secondary Outcome: 24 VAX-24 Pneumococcal Serotype-specific IgG Geometric Mean Concentration (GMCs)
Description: The change from baseline to 1 month post-vaccination in the immune response directed against each of the 24 serotypes was evaluated by measuring IgG levels using an IgG multiplexed electrochemoluminescent assay (ECLA). Values below the lower limit of quantitation (LLOQ) were analyzed as 0.5*LLOQ. Values above the upper limit of quantitation (ULOQ) were analyzed as 1*ULOQ.
Time Frame: 1 month after vaccination
Population: Immunogenicity evaluable population including all participants as treated.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
Number analyzed (Participants) | 48 | 47 | 48 | 45
mcg/mL
  1 | 4.85 [3.24 to 7.26] | 5.36 [3.56 to 8.06] | 4.13 [2.73 to 6.25] | 4.14 [2.71 to 6.34]
  2 | 13.42 [8.97 to 20.07] | 19.04 [12.65 to 28.65] | 9.20 [6.08 to 13.93] | 1.59 [1.04 to 2.44]
  3 | 0.56 [0.37 to 0.84] | 0.64 [0.42 to 0.97] | 0.85 [0.56 to 1.29] | 0.68 [0.44 to 1.04]
  4 | 2.51 [1.60 to 3.95] | 2.50 [1.58 to 3.96] | 2.24 [1.40 to 3.57] | 2.16 [1.34 to 3.48]
  5 | 2.39 [1.44 to 3.96] | 3.20 [1.91 to 5.34] | 2.03 [1.21 to 3.42] | 2.67 [1.57 to 4.56]
  6A | 5.26 [2.97 to 9.34] | 8.61 [4.81 to 15.40] | 6.86 [3.80 to 12.37] | 4.61 [2.52 to 8.44]
  6B | 3.17 [1.78 to 5.65] | 7.50 [4.18 to 13.46] | 5.92 [3.27 to 10.72] | 1.99 [1.08 to 3.66]
  7F | 4.88 [3.25 to 7.35] | 5.50 [3.64 to 8.33] | 7.67 [5.04 to 11.67] | 4.52 [2.94 to 6.96]
  8 | 7.21 [4.66 to 11.16] | 8.08 [5.19 to 12.58] | 5.53 [3.53 to 8.66] | 5.16 [3.25 to 8.17]
  9N | 7.93 [5.68 to 11.06] | 9.83 [7.01 to 13.78] | 8.32 [5.90 to 11.72] | 3.22 [2.27 to 4.58]
  9V | 4.91 [3.11 to 7.75] | 5.56 [3.50 to 8.83] | 7.63 [4.78 to 12.20] | 3.46 [2.14 to 5.60]
  10A | 7.77 [4.63 to 13.03] | 12.31 [7.28 to 20.80] | 9.48 [5.57 to 16.14] | 9.43 [5.46 to 16.27]
  11A | 5.33 [3.67 to 7.73] | 5.46 [3.75 to 7.97] | 5.73 [3.91 to 8.40] | 4.70 [3.18 to 6.96]
  12F | 1.86 [1.17 to 2.95] | 2.77 [1.74 to 4.42] | 2.07 [1.29 to 3.33] | 0.88 [0.54 to 1.42]
  14: number analyzed (Participants) | 48 | 47 | 47 | 45
  14 | 7.93 [4.71 to 13.33] | 12.21 [7.20 to 20.69] | 10.41 [6.08 to 17.81] | 9.08 [5.25 to 15.73]
  15B | 12.16 [7.69 to 19.23] | 17.82 [11.20 to 28.37] | 13.82 [8.63 to 22.14] | 12.48 [7.69 to 20.23]
  17F | 10.81 [7.18 to 16.28] | 10.82 [7.14 to 16.40] | 10.78 [7.07 to 16.43] | 0.56 [0.36 to 0.86]
  18C | 8.17 [4.94 to 13.53] | 11.92 [7.15 to 19.88] | 15.03 [8.95 to 25.23] | 8.25 [4.85 to 14.04]
  19A | 10.58 [6.96 to 16.07] | 13.97 [9.14 to 21.37] | 13.37 [8.69 to 20.57] | 7.84 [5.04 to 12.19]
  19F | 8.21 [4.96 to 13.61] | 9.61 [5.76 to 16.04] | 11.51 [6.85 to 19.34] | 3.14 [1.84 to 5.35]
  20B | 18.18 [13.27 to 24.90] | 24.61 [17.88 to 33.88] | 19.51 [14.12 to 26.98] | 4.77 [3.42 to 6.65]
  22F | 3.26 [2.22 to 4.79] | 6.53 [4.42 to 9.64] | 4.14 [2.79 to 6.14] | 7.99 [5.33 to 11.98]
  23F: number analyzed (Participants) | 47 | 47 | 48 | 45
  23F | 5.16 [3.23 to 8.22] | 9.10 [5.69 to 14.56] | 7.10 [4.41 to 11.44] | 5.31 [3.26 to 8.66]
  33F | 11.96 [8.28 to 17.28] | 14.34 [9.87 to 20.84] | 13.24 [9.07 to 19.34] | 10.82 [7.34 to 15.96]

ADVERSE EVENTS:
Time Frame: 6 months from vaccination
Groups:
- VAX-24 Low Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose level.
  24-Valent Pneumococcal Conjugate Vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose level.
  24-Valent Pneumococcal Conjugate Vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mixed Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg/4.4 mcg dose levels.
  24-Valent Pneumococcal Conjugate Vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20Group 4
All-Cause Mortality (participants affected / at risk) | 0/52 | 1/51 | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/51 | 1/53 | 0/50
Other Adverse Events (participants affected / at risk) | 26/52 | 35/51 | 23/53 | 27/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAX-24 Low Dose (N=52) | VAX-24 Mid Dose (N=51) | VAX-24 Mixed Dose (N=53) | PCV20Group 4 (N=50)
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAX-24 Low Dose (N=52) | VAX-24 Mid Dose (N=51) | VAX-24 Mixed Dose (N=53) | PCV20Group 4 (N=50)
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 5
Pain (Local) (Skin and subcutaneous tissue disorders) | 20 | 32 | 20 | 24
Edema (local) (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 3
Fatigue (General disorders) | 14 | 16 | 8 | 7
Headache (General disorders) | 9 | 6 | 6 | 8
Muscle Pain (Musculoskeletal and connective tissue disorders) | 10 | 14 | 9 | 16
Joint pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3 | 2

LIMITATIONS AND CAVEATS:
Some limitations of this clinical study include the lack of a group, such as 3·3 µg or 4·4 µg, for all serotypes, aimed at understanding whether the dose response of polysaccharide can overcome carrier suppression. The relatively low ethnic diversity of participants is also a limitation, and the sample size was relatively small, both of which will be addressed in larger phase 3 clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall review within the ninety (90) day period. Upon receiving any notification from Sponsor requesting deletion of Confidential Information, correction of inaccuracies, or a delay in publication to allow the filing of patent application, Institution or Investigator shall take the requested action of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT05297578/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT05297578/SAP_002.pdf